CLINICAL TRIAL: NCT03467061
Title: The Effect of Dietary Nitrate on the Oral Microbiota, Markers of Nitric Oxide Bioavailability and Cardiovascular Health in in Young and Older Adults
Brief Title: The Effect of Dietary Nitrate on the Oral Microbiome
Acronym: Microbio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1718/14
Record Dates: First submitted 2017-12-19; First posted 2018-03-15 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Cardiovascular Health; Identify Oral Bacteria Responsible for Nitrate Reduction
MeSH Terms: interventions — Mouthwashes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nitrate-rich beetroot juice (Active Comparator): 2 x 70mL concentrated juice per day for 14 days
  Interventions: Dietary Supplement: Nitrate-rich beetroot juice
- Nitrate-depleted beetroot juice (Placebo Comparator): 2 x 70mL concentrated juice per day for 14 days
  Interventions: Dietary Supplement: Nitrate-depleted beetroot juice
- Antibacterial mouthwash (Other): 2 x 10mL antibacterial mouthwash per day for 14 days
  Interventions: Other: Mouthwash

INTERVENTIONS:
Dietary Supplement: Nitrate-rich beetroot juice — concentrated beetroot juice
  Arms: Nitrate-rich beetroot juice
Dietary Supplement: Nitrate-depleted beetroot juice — concentrated beetroot juice
  Arms: Nitrate-depleted beetroot juice
Other: Mouthwash — 2 x 10 mL antibacterial mouthwash per day for 14 days
  Arms: Antibacterial mouthwash

SUMMARY:
This study evaluates whether dietary manipulation of the oral microbiota modulates cardiovascular health through effects on nitric oxide bioavailability.

DETAILED DESCRIPTION:
Nitric oxide is an important molecule for human health because it controls blood flow and blood pressure. With aging, our ability to make nitric oxide gets worse and our blood pressure tends to increase. We can help the body produce more nitric oxide by supplementing the diet with vegetables, such as beetroot juice, which contains high amounts of nitrate. This has been shown to improve blood flow and blood pressure. The bacteria inside our mouths play an important role in helping convert the ingested nitrate to nitric oxide. The reason for this study is to find out whether there are differences in oral bacteria between young and older adults, and how the oral bacterial community and blood flow and blood pressure might change when diet is supplemented with natural, nitrate-rich beetroot juice and when we use antibacterial mouthwash. This study will help us understand how the bacteria inside our mouths might be useful for keeping us healthy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young (18-30 yr) and older adults (65-80 yr)
* Male and female
* Willing to undergo the experiments as detailed in the informed consent documentation
* Willing and capable of providing written, informed consent.

Exclusion Criteria:

* Individuals receiving medication for pulmonary, cardiovascular, or metabolic conditions, ulcerative colitis or renal disease
* Having an active oral disease or dentures
* Having resting BP >140/90 mmHg
* Having used antibiotics within 3 months
* Lacking willingness or capacity to give informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2021-05-06 (Actual)

PRIMARY OUTCOMES:
Quantity of nitrate -reducing bacteria | 14 days
  Change in total quantity of nitrate-reducing bacteria as measured by sequencing bacterial 16S rRNA genes

SECONDARY OUTCOMES:
Nitric oxide bioavailability - plasma nitrite | 14 days
  Change in nitrite concentration of plasma as measured by ozone-based chemiluminescence
Nitric oxide bioavailability - salivary nitrite | 14 days
  Change in nitrite concentration of saliva as measured by ozone-based chemiluminescence
Nitric oxide bioavailability - plasma nitrate | 14 days
  Change in nitrate concentration of plasma as measured by ozone-based chemiluminescence
Nitric oxide bioavailability - salivary nitrate | 14 days
  Change in nitrate concentration of saliva as measured by ozone-based chemiluminescence
Blood pressure | 14 days
  Change in systolic and diastolic BP
Flow mediated dilation | 14 days
  Change in flow mediated dilation

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Jones, PhD, Principal Investigator — University of Exeter
Locations (1):
- Diabetes & Vascular Medicine Research Centre, Clinical Research Facility, Exeter, Devon, United Kingdom